CLINICAL TRIAL: NCT05012579
Title: A Study of Safety and Efficacy of Transcutaneous Afferent Patterned Stimulation (TAPS) for Reduction of Action Tremor in Parkinson's Disease (PD)
Brief Title: Transcutaneous Afferent Patterned Stimulation (TAPS) for Reduction of Parkinson's Disease (PD) Related Action Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cala Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-02
Record Dates: First submitted 2021-08-03; First posted 2021-08-19 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TAPS delivered by Cala device (Experimental): Two 40-minute TAPS sessions daily for 28 days, recommended as once in the morning and once in the evening.
  Interventions: Device: Cala Device

INTERVENTIONS:
Device: Cala Device — transcutaneous afferent patterned stimulation (TAPS)

SUMMARY:
Demonstrate safety and efficacy of TAPS delivered by a Cala device as a treatment for action tremor in subjects with Parkinson's disease hand tremor

DETAILED DESCRIPTION:
40 patients with PD with at least mild postural tremor were enrolled in a four-week, prospective, single-arm, open-label study of twice daily TAPS therapy. Due to the COVID-19 pandemic, TAPS devices were shipped to patients to run the study remotely. Unsupervised motion assessments were captured at home, and at the beginning and end of the four weeks by telemedicine.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥22 years of age
* Competent and willing to provide written, informed consent to participate in the study
* Clinically significant postural tremor as defined by:

  * Dominant hand/arm exhibiting postural tremor ≥ 2 (while in the off state) as assessed by the MDS-UPDRS postural tremor score
* Stable dose of Parkinson's disease medications, if applicable, for 30 days prior to study entry
* Willing to comply with study protocol requirements including:

  * Having the ability to do telemedicine or video calls for study visits
  * remaining on a stable dosage of Parkinson's medications, if applicable, during the duration of the study
  * no significant caffeine consumption within 8 hours of study visits

Exclusion Criteria:

* Implanted electrical medical device, such as a pacemaker, defibrillator, or deep brain stimulator
* Suspected or diagnosed epilepsy or other seizure disorder
* Swollen, infected, inflamed areas, or skin eruptions, open wounds, or cancerous lesions of skin at stimulation site
* Peripheral neuropathy affecting the tested upper extremity
* Presence of any other neurodegenerative disease or dementia. These may include: multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and Alzheimer's disease.
* Botulinum toxin injection for hand tremor within 6 months prior to study enrollment
* Are participating or have participated in another interventional clinical trial in the last 30 days which may confound the results of this study, unless approved by the Sponsor
* Significant caffeine consumption within 8 hours of study enrollment, which may confound the results of the study, where significant caffeine is considered more than 95 mg (equivalent to a cup of coffee).
* Subjects unable to communicate with the investigator and staff
* Any health condition that in the investigator's opinion should preclude participation in this study
* Pregnancy or anticipated pregnancy during the course of the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cala Clinic, Burlingame, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAPS Delivered by Cala Device
Started | 40
Completed | 37
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: 40 enrolled subjects with PD
Arm/Group | TAPS Delivered by Cala Device
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 6
  Race: African American | 1
  Race: Caucasian | 33

OUTCOME MEASURES:

1. Primary Outcome: Tremor Power
Description: Pre-specified effectiveness endpoints included improvements in (1) objective postural tremor power (primary outcome; assessed using an accelerometer on the device under standard of care medication state at home).
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage of tremor power reduction
Groups:
- Single Arm - TAPS Delivered by Cala Device: Two 40-minute TAPS sessions daily for 28 days, recommended as once in the morning and once in the evening.
  Cala Device: transcutaneous afferent patterned stimulation (TAPS)
Arm/Group | Single Arm - TAPS Delivered by Cala Device
Number analyzed (Participants) | 36
Percentage of tremor power reduction | 64 [54 to 79]

2. Secondary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
Description: Improvement of clinician-ratings of Movement Disorder Society Unified PD Rating Scale (MDS-UPDRS) Part III [Goetz, C.G. et al. Wiley Intersci. 2008] (co-secondary; in medication-off state). Clinician rated patients' tremor pre and post therapy on a scale of 0-4. 0=Normal (no tremor), 4=Severe.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm - TAPS Delivered by Cala Device
Number analyzed (Participants) | 36
units on a scale | 0.6 (0.5)

3. Secondary Outcome: Bain and Findley Activities of Daily Living (BF-ADL)
Description: Improvement of patient-ratings of the Bain and Findley Activities of Daily Living (BF-ADL) [Bain PG, et al. Journal of Neurol, Neuros & Psych 1993] (co-secondary; in medication-off state). Patients' rated ability to perform specific activities pre and post therapy on a scale from 1-4. 1=Able to do the activity without difficulty, 4=Cannot do the activity by yourself.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm - TAPS Delivered by Cala Device
Number analyzed (Participants) | 36
units on a scale | 0.5 (0.5)

4. Secondary Outcome: Percentage of Patients With Clinician and Patient Global Impressions of Improvement Rated < 4 (CGI-I, PGI-I)
Description: Clinician and Patient global impressions of improvement (CGI-I, PGI-I; exploratory) post therapy. This is a rated scale from 1-7, with 1=Very Much Improved to 7=Very Much Worse. Percentage of patients with ratings < 4 (including very much improved, much improved and improved) were computed respectively for CGI-I and PGI-I.
Time Frame: 4 weeks
Measure: Number; unit: percentage of patients with improvement
Arm/Group | Single Arm - TAPS Delivered by Cala Device
Number analyzed (Participants) | 36
percentage of patients with improvement
  PGI-I | 80
  CGI-I | 77

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | TAPS Delivered by Cala Device
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 8/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAPS Delivered by Cala Device (N=40)
Unsteady gait (General disorders) | 1
sore/lesion (Skin and subcutaneous tissue disorders) | 2 — sore/lesion observed in 2 subjects, on the dominant wrist
significant and persistent skin irritation (Skin and subcutaneous tissue disorders) | 1
persistent pain from stimulation (Musculoskeletal and connective tissue disorders) | 1 — pain felt in thumb of treatment hand
significant discomfort with stimulation (General disorders) | 1
twitching of ring finger (Musculoskeletal and connective tissue disorders) | 1 — ring finger on treatment hand
anxiety/insomnia/worsening of tremor at night (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT05012579/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT05012579/SAP_001.pdf